CLINICAL TRIAL: NCT02765854
Title: Phase II Trial of Ixazomib and Dexamethasone Versus Ixazomib, Dexamethasone and Lenalidomide, Randomized With NFKB2 Rearrangement. (Proteasome Inhibitor NFKB2 Rearrangement Driven Trial, PINR)
Brief Title: Ixazomib and Dexamethasone Versus Ixazomib, Dexamethasone and Lenalidomide, Randomized With NFKB2 Rearrangement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Multiple Myeloma Research Consortium (Network); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leon Bernal-Mizrachi, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00077815; NCI-2016-00043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MMRC060 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: Yes

ARMS (3):
- Arm B (ixazomib and dexamethasone) (Experimental): MUTATED NFKB2 REARRANGEMENT: Patients receive ixazomib and dexamethasone as in arm A.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib
- Arm C (ixazomib, dexamethasone, lenalidomide) (Experimental): MUTATED NFKB2 REARRANGEMENT: Patients receive ixazomib and dexamethasone as in arm A and lenalidomide PO daily on days 1-21.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib; Drug: Lenalidomide
- Arm A (ixazomib and dexamethasone) (Active Comparator): UNMUTATED NFKB2 REARRANGEMENT: Patients receive ixazomib and dexamethasone.
  Interventions: Drug: Dexamethasone; Drug: Ixazomib

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Decadron; DexPak; Dexasone; Baycadron; Zema; Diodex; Hexadrol; Maxidex
Drug: Ixazomib — Given PO
  Other Names: MLN9708; Ninlaro; Ixazomib citrate
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; Revlimid
  Arms: Arm C (ixazomib, dexamethasone, lenalidomide)

SUMMARY:
This randomized phase II trial studies how well ixazomib and dexamethasone or ixazomib, dexamethasone, and lenalidomide work based on the presence of the rearrangement of a gene called nuclear factor of kappa light polypeptide gene enhancer in B-cells 2 (NFKB2) in treating patients with multiple myeloma that has returned after a period of improvement or does not respond to treatment. Ixazomib may stop the growth of cancer cells by blocking enzymes called proteasomes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lenalidomide may stimulate the immune system against cancer cells and may also prevent the growth of new blood vessels that tumors need to grow. It is not yet known whether ixazomib and dexamethasone, or ixazomib, dexamethasone, and lenalidomide are more effective in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To test whether the NFKB2 rearrangement can guide the selection of treatment (ixazomib [ixazomib citrate] plus dexamethasone [Id] or ixazomib plus lenalidomide and dexamethasone [IRd]) by conducting the following comparisons:

I. To compare the response rate at 4 cycles between patients treated with Id and patients treated with IRd and confirm the lack of significant difference in overall response.

II. To compare the response rate at 4 cycles between non-rearranged and rearranged NFKB2 treated with Id and confirm that NFKB2 rearrangement is associated with reduce response rate.

III. To compare the responses rate at 4 cycles of patients with rearranged NFKB2 treated with Id or IRd and confirm that adding lenalidomide increases the response rate in this population.

SECONDARY OBJECTIVES:

I. To determine time to treatment failure (TTF).

II. To determine the frequency and severity of adverse events (AE) in IRd treated cohort.

III. To identify novel transcribed mutations associated with Id and IRd resistance in patients with multiple myeloma (MM).

IV. To determine the prevalence of NFKB2 rearrangement in relapsed/refractory MM patients screened in the study.

V. To determine the prevalence of NFKB2 rearrangement according to the type of previous therapies received in all patients screened in the study.

VI. To determine the toxicity profile of the study drugs according to the presence of NFKB2 rearrangement.

VII. Delineate transcribed mutations associated with relapse or refractoriness to Id or IRd treatment by ribonucleic acid (RNA)-sequencing.

OUTLINE:

ARM A (UNMUTATED NFKB2 REARRANGEMENT): Patients receive ixazomib orally (PO) on days 1, 8, and 15 and dexamethasone PO on days 1, 8, 15, and 22.

Patients with mutated NFKB2 rearrangement are randomized in to 1 of 2 treatment arms.

ARM B (MUTATED NFKB2 REARRANGEMENT): Patients receive ixazomib and dexamethasone as in arm A.

ARM C (MUTATED NFKB2 REARRANGEMENT): Patients receive ixazomib and dexamethasone as in arm A and lenalidomide PO daily on days 1-21.

In all arms, cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients may proceed to autologous stem cell transplant after 4 cycles of treatment.

After completion of study, patients are followed up monthly.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care
* Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International Units (mIU)/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and ixazomib and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide through 90 days after the last dose of study drug; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy from the time of signing the informed consent form through 90 days after the last dose of study drug; in the event that the male patients choose to agree to practice true abstinence, this must follow the timelines detailed above; all patients assigned to the lenalidomide treatment group must be registered in and must comply with all requirements of the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program

  * *A female of childbearing potential is a sexually mature woman who:

    * 1) has not undergone a hysterectomy or bilateral oophorectomy; or
    * 2) has not been naturally postmenopausal for at least 24 consecutive months
* Multiple myeloma diagnosed according to standard criteria either currently or at the time of initial diagnosis
* The patient has confirmed relapsed or refractory MM
* For patients that relapse following a response to prior treatment with bortezomib or carfilzomib, six months must have elapsed since the last dose of treatment
* The patient has received 1 to 3 prior lines of therapy. By definition, a single line of therapy may consist of 1 or more agents, and may include induction, hematopoietic stem cell transplantation, and maintenance therapy. Radiotherapy, bisphosphonate, or a single short course of steroids (ie, less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days) would not be considered prior lines of therapy
* Patients must have measurable disease defined by at least 1 of the following measurements:

  * Serum M-protein ≥ 1.0 g/dL (≥ 10 g/L) for an immunoglobulin (Ig)G myeloma, ≥ 0.1 g/dL for an immunoglobulin D (IgD) myeloma or 0.5 g/dL (≥ 5g/L) for an immunoglobulin A (IgA) myeloma
  * Urine light chain ≥ 200 mg/24 hours
  * Serum free light chain ≥ 10 mg/dL provided the free light chain (FLC) ratio is abnormal
  * Patients with oligo- or non-secretory disease must have bone marrow involvement with at least 30% plasmacytosis on aspiration
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2
* Absolute neutrophil count (ANC) ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³; in the case that platelets are between 50,000-75,000, the patient can be enrolled if the plasma cell count in the bone marrow is superior to ≥ 50%; to meet this hematological eligibility no transfusion support and hematological growth factor are not allowed within 7 days before study enrollment
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Serum creatinine ≤ 2.5 mg/dL or a calculated creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* The patient is refractory to carfilzomib or bortezomib; (refractory is defined as patients who never achieved a response and progressed while on carfilzomib or bortezomib or within 60 days of completing treatment)
* Prior treatment with any investigational proteasome inhibitor within 6 months of study entry
* Female patients who are breast feeding or have a positive serum pregnancy test during the screening period
* Failure to have fully recovered (ie, > grade 1 toxicity) from the reversible effects of prior chemotherapy
* Diarrhea > grade 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03
* Prior chemotherapy and/or immunotherapy within 14 days before enrollment; major surgery within 14 days before enrollment and minor surgery within 7 days prior to cycle 1 day 1
* Radiotherapy within 14 days before enrollment; if the involved field covered ≤ 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy
* Central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort
* Active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially compromise the patient's ability to understand the patient information, to give informed consent, to comply with the treatment according to this protocol or complete the study
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Patient has ≥ grade 2 peripheral neuropathy or neuropathy with pain, regardless of grade that is seen on clinical examination during the screening period
* Known intolerance to immunomodulatory drugs (IMiDs)
* History of allergic reaction/hypersensitivity to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or lenalidomide, including difficulty swallowing
* Participation in other clinical trials, including those with other investigational agents not included in this trial, such as monoclonal antibodies, within 30 days of the start of this trial and throughout the duration of this trial
* Corticosteroid doses > 10 mg/day of prednisone or equivalent within 14 days prior to cycle 1 day 1
* Autologous or allogeneic stem cell or bone marrow transplant within 3 months prior to cycle 1 day 1
* Cytotoxic therapy within 21 days prior to cycle 1 day (D) 1
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Bernal-Mizrachi, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Michigan/Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University/Siteman Cancer Center, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Started | 22 | 21 | 27
Completed | 22 | 21 | 27
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone) | Total
Number analyzed (Participants) | 22 | 21 | 27 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 12 | 26
  >=65 years | 15 | 14 | 15 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 14 | 30
  Male | 16 | 11 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 13 | 29
  White | 12 | 13 | 13 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 27 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is to Test Whether the NFKB2 Rearrangement Can Guide the Selection of Treatment (Ixazomib Plus Dexamethasone (Id) or Ixazomib Plus Lenalidomide and Dexamethasone (IRd)) by Conducting the 3 Following Comparisons
Description: Comparison to a historical control: The overall response rate (ORR) of each arm at 4 cycles (112 days) is compared to the historical RR of 30%. Arm A or Arm C is designed to detect an improved RR of 60% vs. 30% using Simon's 2-stage Optimum design with a power of at least 90% and an alpha error of 5%., respectively. For Arm B will achieve a power of at least 80% at the significance level of 0.05 to claim that Arm B has equivalent RR as the historical RR of 30% assuming an equivalence tolerance of +/- 20% when the true RR of Arm B is approximately 30%.
  Response Rate is defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 112 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Number analyzed (Participants) | 22 | 21 | 27
Participants
  Yes: Response Achieved at Four Cycles | 8 | 14 | 16
  No: Response Achieved at Four Cycles | 14 | 7 | 11

2. Secondary Outcome: Time to Treatment Failure
Description: Kaplan-Meier curves will be used for the time to treatment failure according to the Arm of treatment utilized. Kaplan-Meyer curve analysis was performed to evaluate the time to treatment failure comparison.
Time Frame: Up to 30 months
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Number analyzed (Participants) | 22 | 21 | 27
Months
  6 Months | 0.495 [0.259 to 0.693] | 0.683 [0.419 to 0.847] | 0.729 [0.512 to 0.861]
  12 Months | 0.353 [0.142 to 0.575] | 0.312 [0.103 to 0.551] | 0.729 [0.512 to 0.861]
  18 Months | 0.283 [0.095 to 0.508] | 0.312 [0.103 to 0.551] | 0.663 [0.425 to 0.821]
  24 Months | 0.141 [0.024 to 0.357] | 0.156 [0.026 to 0.388] | 0.505 [0.249 to 0.715]
  30 Months | 0.141 [0.024 to 0.357] | 0.078 [0.005 to 0.294] | 0.421 [0.176 to 0.65]

3. Secondary Outcome: Prevalence of NFKB2 Rearrangement in Relapsed/Refractory Multiple Myeloma Patients Screened in the Study.
Description: To determine the prevalence of NFKB2 rearrangement according to the type of previous therapies received in all patients screened in the study.
Time Frame: At baseline and month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Number analyzed (Participants) | 22 | 21 | 27
Participants | 22 | 21 | 0

4. Secondary Outcome: Percentage of Patients With Response at Baseline and at 12 Months
Description: Determine percentage of patients with response at 8 cycles of treatment
Time Frame: At baseline and at 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Number analyzed (Participants) | 22 | 21 | 27
percentage of participants
  Baseline | 31 | 42 | 37
  Month 12 | 35 | 35 | 73

5. Secondary Outcome: Incidence of Adverse Events
Description: Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity. Additional safety analyses may be performed to most clearly enumerate rates of toxicities and to further define the safety profile of Id or IRd combinations. Treatment-emergent events will be tabulated.
Time Frame: 30 days post-treatment, up to a total of 1 year
Measure: Number; unit: participants
Arm/Group | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) | Arm A (Ixazomib and Dexamethasone)
Number analyzed (Participants) | 22 | 21 | 27
participants
  Agitation | 0 | 0 | 1
  Altered Mental Status | 0 | 0 | 1
  Anemia | 1 | 1 | 1
  Anxiety | 0 | 1 | 0
  Ari | 1 | 0 | 0
  Bone Pain | 4 | 1 | 0
  Bp195/90 | 0 | 0 | 1
  Cardiopulmonary Arrest, Presumed | 0 | 0 | 1
  Cellulitis | 1 | 0 | 0
  Colitis | 0 | 1 | 4
  Conjunctivitis | 4 | 0 | 2
  Constipation | 0 | 1 | 0
  Death-Multisystem Organ Failure | 0 | 0 | 1
  Dehydration | 0 | 1 | 0
  Diarrhea | 0 | 1 | 2
  Dress Syndrome | 0 | 1 | 0
  Dysphagia | 0 | 0 | 2
  Ecchymosis | 1 | 0 | 0
  Edema | 0 | 0 | 1
  Fatigue | 1 | 0 | 1
  Gastrointestinal Bleed | 0 | 0 | 1
  Generalized Weakness | 0 | 0 | 1
  Hepatitis | 0 | 0 | 1
  Hernia | 0 | 1 | 0
  Hyperglycemia | 0 | 2 | 0
  Hypertension | 0 | 1 | 1
  Hyponatremia | 0 | 0 | 1
  Hypophosphatemia | 0 | 1 | 0
  Insomnia | 0 | 0 | 1
  Leucopenia | 0 | 1 | 0
  Lymphopenia | 0 | 0 | 1
  Nausea And Vomiting | 0 | 0 | 1
  Neuropathy | 0 | 3 | 2
  Neutropenia | 0 | 2 | 0
  Neutropenic Fever | 0 | 1 | 0
  Pancytopenia | 0 | 1 | 0
  Pedestrian In Motor Vehicle Accident | 0 | 0 | 1
  Pneumonia | 3 | 3 | 6
  Rash | 0 | 1 | 1
  Sepsis | 0 | 0 | 1
  Sinus Tachycardia | 0 | 0 | 1
  Supraventricular Tachycardia | 0 | 1 | 0
  Thrombocytopenia | 0 | 6 | 2
  Tremors | 0 | 1 | 0
  Tumor Lysis Syndrome | 0 | 0 | 1
  Upper Respiratory Infection | 0 | 0 | 6
  Urinary Tract Infection | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm A (Ixazomib and Dexamethasone) | Arm B (Ixazomib and Dexamethasone) | Arm C (Ixazomib, Dexamethasone, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 20/27 | 10/22 | 10/21
Other Adverse Events (participants affected / at risk) | 20/27 | 10/22 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Ixazomib and Dexamethasone) (N=27) | Arm B (Ixazomib and Dexamethasone) (N=22) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) (N=21)
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — suspected myocardial infarction.
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — presumed
cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Conjunctivtis (Eye disorders) | 0 (0) | 4 (4) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) — Multisystem Organ Failure
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dress Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MVA (General disorders) | 1 (1) | 0 (0) | 0 (0) — Pedestrian in Motor Vehicle Accident
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Suspected Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — negative blood culture
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Ixazomib and Dexamethasone) (N=27) | Arm B (Ixazomib and Dexamethasone) (N=22) | Arm C (Ixazomib, Dexamethasone, Lenalidomide) (N=21)
Agitation (Psychiatric disorders) | 1 | 0 | 0
Altered Mental Status (General disorders) | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Cardiopulmonary Arrest, Presumed (Cardiac disorders) | 2 | 0 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 6 | 0 | 2
Conjunctivits (Eye disorders) | 2 | 8 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 0 | 1
Dress Syndrome (General disorders) | 0 | 0 | 2
Dysphagia (Nervous system disorders) | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Edema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0
Gastrointestinal Bleed (Gastrointestinal disorders) | 2 | 0 | 0
Generalized Weakness (General disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hernia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphopenia (General disorders) | 1 | 0 | 0
Nausea And Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Neuropathy (Nervous system disorders) | 2 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 4
Neutropenic Fever (General disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pedestrian In Motor Vehicle Accident (General disorders) | 2 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Sepsis; Negative Blood Cultures (Infections and infestations) | 2 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 9
Tremors (Nervous system disorders) | 0 | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 2 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 6 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02765854/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02765854/ICF_000.pdf